CLINICAL TRIAL: NCT01317680
Title: Low Intensity Shock Wave Therapy for Erectile Dysfunction in Post Radical Prostatectomy Patients Not Responding to PDE5 Inhibitors- a Double Blind Placebo Controlled Study (LI-ESWT)
Brief Title: Low Intensity Shock Wave Therapy (LI-ESWT) for Erectile Dysfunction in Post Radical Prostatectomy Patients Not Responding to PDE5 Inhibitors (LI-ESWT)
Acronym: LI-ESWT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, i_gruenwald, MD, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0037-11-RMB
Record Dates: First submitted 2011-03-08; First posted 2011-03-17 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; ED; PDE5 inhibitors; LI-ESWT
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment LI-ESWT (Active Comparator): Device: Extracorporeal Shockwave Therapy Generator (Omnispec model ED1000) Gel is spread around the penis and on the Shock Wave applicator and Treatment (12 sessions in total) of 300 shocks per site, on 5 penile anatomical sites.
  Interventions: Device: Omnispec model ED1000
- Sham control (Placebo Comparator): We use the same probe that induces the same sensation on the penis and the same noise yet no energy.
  Interventions: Device: Sham control

INTERVENTIONS:
Device: Omnispec model ED1000 — Device: Extracorporeal Shockwave Therapy Generator (Omnispec model ED1000) Gel is spread around the penis and on the Shock Wave applicator and Treatment (12 sessions in total) of 300 shocks per site, on 5 penile anatomical sites.
  Arms: Treatment LI-ESWT
Device: Sham control — We use the same probe that induces the same sensation on the penis and the same noise yet no energy
  Arms: Sham control

SUMMARY:
Low intensity shock waves (LISW) have been proven in animal studies to induce local growth of new blood vessels. The investigators hypothesized that LISW therapy could improve the symptoms of patients with erectile dysfunction resulting from a problem of blood supply (damage that can occur after radical prostatectomy in addition to neural damage or solely) that do not respond to oral therapy (PDE-5 inhibitors).

ELIGIBILITY:
Inclusion Criteria:

* Prior prostatectomy surgery
* ED of more than 6 months
* Rigidity score < 3 during PDE5i therapy
* Non- hormonal, neurological or psychological pathology Stable heterosexual relationship for more than 3 months

Exclusion Criteria:

* Any unstable medical, psychiatric, spinal cord injury and penile anatomical abnormalities
* Clinically significant chronic hematological disease
* Anti-androgens, oral or injectable androgens
* Radiotherapy in pelvic region

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-03 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Increase in IIEF ED Domain Questionaire of >5 is considered as a treatment success | 3 months

SECONDARY OUTCOMES:
Rigidity Score Questionaire- an increase of at least 1 point is considered as a treatment success | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Center, Haifa, Israel